CLINICAL TRIAL: NCT00291915
Title: Methotrexate Alone Versus Methotrexate in Combination With Adalimumab in Early Arthritis
Brief Title: Multicenter Randomized Prospective Trial Comparing Methotrexate Alone or in Combination With Adalimumab in Early Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goupe d'Etudes et de Recherche Clinique En Rhumatologie (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUEPARD-GERCER 2122
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2006-02-15 (Estimated); Status verified 2006-02

CONDITIONS: Rheumatoid Arthritis; Arthritis
Keywords: early arthritis, methotrexate, adalimumab
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Adalimumab; Methotrexate

INTERVENTIONS:
Drug: Adalimumab
Drug: Methotrexate

SUMMARY:
Evaluation of two treatment modalities in early potentially severe early arthritis ( Methotrexate alone or in combination with adalimumab)

DETAILED DESCRIPTION:
Patients: early ( less than 6 months), active ( DAS>5.2),potentially severe ( Leiden score>6) Study design:12 months, prospective , randomized, open Study treatments: Methotrexate at a weekly dose of 0.3mg/kilo alone or in combination with adalimumab 40 mg every the other week Outcome measures: DAS over the 12 months

ELIGIBILITY:
Inclusion Criteria:

* Early Active Potentially severe arthritis

Exclusion Criteria:

* contra indication of methotrexate or anti TNF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-05; Study Completion 2007-03

PRIMARY OUTCOMES:
Disease Activity Score

SECONDARY OUTCOMES:
-Radiological score
-Functional impairment ( HAQ)
-Pain (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Maxime DOUGADOS, MD, Principal Investigator — Hopital Cochin Paris FRance
Locations (1):
- Hopital Cochin, Paris, France